CLINICAL TRIAL: NCT02649660
Title: Lipidomics and Functional Analyses of Platelets in Fabry Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Spital Linth (Other Government)
Collaborators: University of Zurich (Other); National University of Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: FabryPlatelets
Record Dates: First submitted 2015-12-06; First posted 2016-01-07 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; Platelets; Lipidomics; Sphingolipids; α-Galactosidase A; Globotriaosylceramide; Gb3; GL-3; CD77; Alpha-galactosidase; Platelet activation; Lysosomal storage disease; LysoGb3; Spingosine-1-Phosphate; Platelet function; CD62P; P-selectin
MeSH Terms: conditions — Fabry Disease; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma, serum and platelet isolates
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to evaluate whether platelets are biochemically and functionally altered in Fabry disease (FD) and therefore possibly implicated in FD manifestations such as cerebrovascular events. To test this hypothesis the investigators aim to compare platelet and plasma lipid profiles, as well as platelet function and coagulation parameters of FD patients and healthy controls.

DETAILED DESCRIPTION:
Fabry disease (FD) is a severe X-linked inborn error of the lysosomal glycosphingolipid metabolism. FD patients have significantly increased risks for cardiac and cerebrovascular events, which can also occur early and in absence of the typical FD symptoms. However, the pathophysiological mechanisms leading to vascular occlusion and ischemia in FD are largely unclear. Prevention of recurrent cerebrovascular events is usually based on empirical anti-platelet therapy.

Prothrombotic states and partially activated platelets have been reported for FD patients. Platelets contain glycosphingolipids, including globotriaosylceramide (Gb3), and have lysosomal α-galactosidase activity. To investigate whether the lack of or the reduced α-galactosidase enzyme activity present in Fabry disease affects platelet lipid metabolism the investigators plan to perform LC-MS-based lipidomics analyses of platelets and plasma in FD patients and healthy controls. To assess whether platelets are functionally altered in FD, the investigators aim to determine the activation status, activability, aggregability and other parameters along with plasma markers of coagulation using flow cytometry, aggregometry and immunoassays.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers: without any known cardiovascular, cerebrovascular and renal diseases and without any known conditions affecting platelet function, blood coagulation and lipid metabolism.
* Patients: Genetically confirmed Fabry Disease
* Adult persons (18-65 years old), both female and male
* Informed written consent

Exclusion Criteria:

* Failure to meet inclusion criteria
* Pregnancy (as declared by the study participant, no pregnancy test will be performed)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Fabry Disease and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in sphingolipid profiles of platelets and plasma between Fabry disease patients and healthy subjects | Baseline
  Determination of sphingolipid concentrations in isolated platelets and plasma by targeted LC-MS (liquid chromatography mass spectrometry)-based lipidomics analysis of globotriaosylceramides (Gb3), globotriaosylspingosines (Lyso-Gb3), globotetraosylceramides (Gb4), lactosylceramides (LacCer), glucosylceramides, ceramides, sphingomyelins, sphingosines and sphingosine-1-phosphates.
Differences in platelet function assessed by aggregometry | Baseline
  Determination of platelet aggregation after agonist stimulation with TRAP (thrombin receptor activator peptide), ADP (adenosine disphosphate) and arachidonic acid by light transmission aggregometry.

SECONDARY OUTCOMES:
Differences in expression of the platelet activation marker P-selectin (CD62P) between Fabry disease patients and healthy subjects at baseline and after agonist stimulation | Baseline
  Flow cytometric analysis of platelet surface expression of CD62P in whole blood determined at baseline and after platelet activation with the agonists TRAP (thrombin receptor activator peptide), ADP, and arachidonic acid.
Differences in expression of the platelet activation marker CD63 between Fabry disease patients and healthy subjects at baseline and after agonist stimulation | Baseline
  Flow cytometric analysis of platelet surface expression of CD63 in whole blood determined at baseline and after platelet activation with the agonists TRAP (thrombin receptor activator peptide), ADP, and arachidonic acid.
Differences in plasma levels of the platelet activation marker soluble P-selectin between Fabry disease patients and healthy subjects | Baseline
  Plasma concentrations of soluble P-selectin (soluble CD62P) are determined by ELISA (enzyme-linked immunosorbent assay)
Differences in plasma levels of the platelet activation marker sCD40L between Fabry disease patients and healthy subjects | Baseline
  Plasma concentrations of sCD40L (soluble CD40 ligand) are determined by ELISA (enzyme-linked immunosorbent assay)
Differences in presence of platelet aggregates between Fabry disease patients and healthy subjects | Baseline
  Flow cytometric assessment of platelet-platelet and platelet-leukocyte aggregates
Differences of alpha-galactosidase A enzyme activity in plasma and isolated platelets between Fabry disease patients and healthy subjects | Baseline
  Analysis of the alpha-galactosidase A enzyme activity using a fluorometric enzyme assay with 4-methylumbelliferyl-α-D-galactopyranoside as substrate.
Differences in phospholipid profiles in platelets and plasma between Fabry disease patients and healthy subjects | Baseline
  Determination of phospholipid concentrations in isolated platelets and plasma by targeted LC-MS-based lipidomics analysis of phosphatidylcholines, phosphatidylserines, phosphatidylinositols, and phosphatidylethanolamines.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alexandre Krayenbühl, MD, Principal Investigator — Spital Linth
Locations (2):
- Switzerland (2):
  - Spital Linth, Uznach, Canton of St. Gallen
  - University Hospital, Zürich, Zurich, Canton of Zurich

REFERENCES:
- [Background] Feldt-Rasmussen U. Fabry disease and early stroke. Stroke Res Treat. 2011;2011:615218. doi: 10.4061/2011/615218. Epub 2011 Jun 23. PMID 21776363
- [Background] Tao RV, Sweeley CC, Jamieson GA. Sphingolipid composition of human platelets. J Lipid Res. 1973 Jan;14(1):16-25. PMID 4701549
- [Background] Beutler E, Kuhl W, Matsumoto F, Pangalis G. Acid hydrolases in leukocytes and platelets of normal subjects and in patients with Gaucher's and Fabry's disease. J Exp Med. 1976 Apr 1;143(4):975-80. doi: 10.1084/jem.143.4.975. PMID 3620
- [Result] Sims K, Politei J, Banikazemi M, Lee P. Stroke in Fabry disease frequently occurs before diagnosis and in the absence of other clinical events: natural history data from the Fabry Registry. Stroke. 2009 Mar;40(3):788-94. doi: 10.1161/STROKEAHA.108.526293. Epub 2009 Jan 15. PMID 19150871
- [Result] Igarashi T, Sakuraba H, Suzuki Y. Activation of platelet function in Fabry's disease. Am J Hematol. 1986 May;22(1):63-7. doi: 10.1002/ajh.2830220110. PMID 3006478
- [Result] DeGraba T, Azhar S, Dignat-George F, Brown E, Boutiere B, Altarescu G, McCarron R, Schiffmann R. Profile of endothelial and leukocyte activation in Fabry patients. Ann Neurol. 2000 Feb;47(2):229-33. PMID 10665494
- [Result] Vedder AC, Biro E, Aerts JM, Nieuwland R, Sturk G, Hollak CE. Plasma markers of coagulation and endothelial activation in Fabry disease: impact of renal impairment. Nephrol Dial Transplant. 2009 Oct;24(10):3074-81. doi: 10.1093/ndt/gfp263. Epub 2009 Jun 10. PMID 19515805